CLINICAL TRIAL: NCT02272816
Title: A Multi-Centre Phase II Study Using Carboplatin AUC-10 for Metastatic Seminoma With IGCCCG Good Prognosis Disease-Therapy Directed by Initial Metabolic Response on PET-CT
Brief Title: Carboplatin AUC-10 With Early PET Scanning in Metastatic Seminoma
Acronym: Car-PET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: University College London Hospitals (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 007065; 2009-009882-33 (EudraCT Number)
Record Dates: First submitted 2012-11-06; First posted 2014-10-23 (Estimated); Results first posted 2019-01-25 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2018-08

CONDITIONS: Metastatic Seminoma
MeSH Terms: conditions — Seminoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Carboplatin AUC-10 (Experimental)
  Interventions: Drug: Carboplatin AUC-10

INTERVENTIONS:
Drug: Carboplatin AUC-10 — Carboplatin AUC-10 according to the Calvert formula [10 x (glomerular filtration rate (ml/min) + 25)]mg given in 5% glucose over 1 hour every 21 days for 3 or 4 cycles.

SUMMARY:
This study evaluated the safety, efficacy and toxicity of carboplatin area under the curve (AUC)-10 in metastatic seminoma to see if, by using fluoro-deoxyglucose (FDG) positron emission tomography-computed tomography (PET-CT) to assess metabolic response, the number of patients requiring 4 cycles can be reduced. Carboplatin AUC-10 was given every 21 days. A PET-CT scan was carried out on day 17-21 of the first cycle. If the PET - CT scan showed a complete response patients received 3 cycles of treatment. If the PET - CT scan did not show a complete response patients received 4 cycles of treatment. After treatment, patients were followed up for 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Metastatic seminoma with International Germ Cell Consensus Classification (IGCCCG) good prognosis.
2. Glomerular filtration rate (GFR) by Ethylenediaminetetraacetic acid (EDTA) clearance over 25 ml/min.
3. Eastern Cooperative Oncology Group (ECOG) Performance status 0-3.
4. Normal Alpha-fetoprotein (All levels of Human chorionic gonadotropin and Lactate dehydrogenase are acceptable).
5. Males aged ≥18 and ≤75 years.
6. Able to give written informed consent prior to study entry.
7. Patients must be sterile or agree to use adequate contraception during the period of therapy.

Exclusion Criteria:

1. Metastatic seminoma with any non-pulmonary visceral metastases.
2. Raised Alpha-fetoprotein.
3. Any previous chemotherapy or radiotherapy.
4. Currently enrolled in any other investigational drug study.
5. Other malignancy except basal cell.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-02-13 (Actual); Primary Completion 2017-10-13 (Actual); Study Completion 2017-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Shamash, MD FRCP, Principal Investigator — Barts & The London NHS Trust
Locations (2):
- United Kingdom (2):
  - Barts Health NHS Trust, London
  - Hillingdon Hospitals NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Horwich A, Oliver RT, Wilkinson PM, Mead GM, Harland SJ, Cullen MH, Roberts JT, Fossa SD, Dearnaley DP, Lallemand E, Stenning SP; MRC Testicular Tumour Working Party. A medical research council randomized trial of single agent carboplatin versus etoposide and cisplatin for advanced metastatic seminoma. MRC Testicular Tumour Working Party. Br J Cancer. 2000 Dec;83(12):1623-9. doi: 10.1054/bjoc.2000.1498. PMID 11104556
- [Background] Bokemeyer C, Kollmannsberger C, Stenning S, Hartmann JT, Horwich A, Clemm C, Gerl A, Meisner C, Ruckerl CP, Schmoll HJ, Kanz L, Oliver T. Metastatic seminoma treated with either single agent carboplatin or cisplatin-based combination chemotherapy: a pooled analysis of two randomised trials. Br J Cancer. 2004 Aug 16;91(4):683-7. doi: 10.1038/sj.bjc.6602020. PMID 15266338
- [Background] Shamash J, McLaren B, LeVay JH, Ong J, Murray P, Asterling S, Oliver RT. Carboplatin AUC8 in combination with etoposide and bleomycin in the treatment of intermediate and poor-risk metastatic germ cell tumours: a phase II study. Cancer Chemother Pharmacol. 2001 Apr;47(4):370-2. doi: 10.1007/s002800000217. PMID 11345655
- [Background] Horwich A, Sleijfer DT, Fossa SD, Kaye SB, Oliver RT, Cullen MH, Mead GM, de Wit R, de Mulder PH, Dearnaley DP, Cook PA, Sylvester RJ, Stenning SP. Randomized trial of bleomycin, etoposide, and cisplatin compared with bleomycin, etoposide, and carboplatin in good-prognosis metastatic nonseminomatous germ cell cancer: a Multiinstitutional Medical Research Council/European Organization for Research and Treatment of Cancer Trial. J Clin Oncol. 1997 May;15(5):1844-52. doi: 10.1200/JCO.1997.15.5.1844. PMID 9164194
- [Background] Gore M, Mainwaring P, A'Hern R, MacFarlane V, Slevin M, Harper P, Osborne R, Mansi J, Blake P, Wiltshaw E, Shepherd J. Randomized trial of dose-intensity with single-agent carboplatin in patients with epithelial ovarian cancer. London Gynaecological Oncology Group. J Clin Oncol. 1998 Jul;16(7):2426-34. doi: 10.1200/JCO.1998.16.7.2426. PMID 9667260
- [Background] Cheson BD, Pfistner B, Juweid ME, Gascoyne RD, Specht L, Horning SJ, Coiffier B, Fisher RI, Hagenbeek A, Zucca E, Rosen ST, Stroobants S, Lister TA, Hoppe RT, Dreyling M, Tobinai K, Vose JM, Connors JM, Federico M, Diehl V; International Harmonization Project on Lymphoma. Revised response criteria for malignant lymphoma. J Clin Oncol. 2007 Feb 10;25(5):579-86. doi: 10.1200/JCO.2006.09.2403. Epub 2007 Jan 22. PMID 17242396
- [Background] Juweid ME, Stroobants S, Hoekstra OS, Mottaghy FM, Dietlein M, Guermazi A, Wiseman GA, Kostakoglu L, Scheidhauer K, Buck A, Naumann R, Spaepen K, Hicks RJ, Weber WA, Reske SN, Schwaiger M, Schwartz LH, Zijlstra JM, Siegel BA, Cheson BD; Imaging Subcommittee of International Harmonization Project in Lymphoma. Use of positron emission tomography for response assessment of lymphoma: consensus of the Imaging Subcommittee of International Harmonization Project in Lymphoma. J Clin Oncol. 2007 Feb 10;25(5):571-8. doi: 10.1200/JCO.2006.08.2305. Epub 2007 Jan 22. PMID 17242397
- [Background] A'Hern RP. Sample size tables for exact single-stage phase II designs. Stat Med. 2001 Mar 30;20(6):859-66. doi: 10.1002/sim.721. PMID 11252008
- [Background] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009
- [Derived] Shamash J, Syed R, Sarker SJ, Sarwar N, Sharma A, Mutsvangwa K, Coetzee C, Wilson P, Rustin GJ. A phase II study of carboplatin AUC-10 guided by positron emission tomography-defined metabolic response in metastatic seminoma. Eur J Cancer. 2019 Jul;115:128-135. doi: 10.1016/j.ejca.2019.04.013. Epub 2019 May 25. PMID 31136925

RESULTS

PARTICIPANT FLOW:
Groups:
- Carboplatin AUC-10: Carboplatin area under the curve (AUC)-10: Carboplatin AUC-10 according to the Calvert formula [10 x (glomerular filtration rate (ml/min) + 25)]mg given in 5% glucose over 1 hour every 21 days for 3 or 4 cycles.
Period: Overall Study
Arm/Group | Carboplatin AUC-10
Started | 48
Completed | 47
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Carboplatin AUC-10
Number analyzed (Participants) | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 47
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 48
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 48
Primary Tumour [Count of Participants; unit: Participants] — Location of primary tumour.
  Participants
    Testis | 46
    Mediastinum | 1
    Retroperitoneum | 1
Sites of Metastases [Count of Participants; unit: Participants] — Count of participants with metastases in specified locations.
  Participants
    Lung | 2
    Lymph node | 29
    Other | 9
    Not recorded | 8
Eastern Cooperative Oncology Group Performance Status (ECOG PS) [Count of Participants; unit: Participants] — A quantification of participants daily living ability. 0. Fully active, able to carry out all normal activity without restriction.
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature
  2. Ambulatory and capable of all self-care, but unable to carry out any work activities. Up and about more than 50% of waking hours.
  3. Capable of only limited self-care. Confined to bed or chair more than 50% of waking hours.
  Participants
    ECOG PS = 0 | 41
    ECOG PS = 1 | 2
    ECOG PS = 2 | 0
    ECOG PS = 3 | 0
    Not recorded | 5
Stage of Disease [Count of Participants; unit: Participants] — Categories of stage 2 cancer:
  2A - Cancer has spread to one or more lymph nodes, but no node is larger than 2 cm.
  2B - Cancer has spread to at least one lymph node, which is between 2 cm and 5 cm in size.
  2C - Cancer has spread to at least one lymph node that is larger than 5 cm.
  N/A - Mediastinal cancer
  Participants
    2A | 13
    2B | 23
    2C | 11
    N/A | 1
Tumour Marker: Alpha-fetoprotein [Count of Participants; unit: Participants]
  Normal | 48
  Elevated | 0
Tumour Marker: Beta-Human Chorionic Gonadotropin [Count of Participants; unit: Participants]
  Normal | 36
  Elevated | 12
Tumour Marker: Lactate Dehydrogenase [Count of Participants; unit: Participants]
  Normal | 34
  Elevated (< 3 x ULN) | 11
  Elevated (≥ 3 x ULN) | 2
  Not recorded | 1
Glomerular Filtration Rate [Count of Participants; unit: Participants] — Ethylenediaminetetraacetic acid (EDTA) clearance (43 participants) or estimated creatinine clearance determined by Cockcroft-Gault equation (5 participants).
  Participants
    25 - 120 ml/min | 35
    > 120 ml/min | 13

OUTCOME MEASURES:

1. Primary Outcome: 2 - Year Progression Free Survival
Description: Number of participants progression free 2 years after registration.
Time Frame: 2 years
Population: All participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Carboplatin AUC-10
Number analyzed (Participants) | 48
Participants | 46
Statistical Analysis 1: Comparison: Carboplatin AUC-10; Test type: Other; Percentage = 95.6, 95% CI 1-sided [upper limit 98.6]

2. Secondary Outcome: Metabolic Response Rate
Description: Number of participants achieving i) complete metabolic response (CR) and ii) partial metabolic response (PR) after one cycle of treatment.
Time Frame: 21 days
Population: All participants who completed one cycle of treatment and underwent PET-CT scan on day 17-21.
Measure: Count of Participants; unit: Participants
Arm/Group | Carboplatin AUC-10
Number analyzed (Participants) | 47
Participants
  CR | 21
  PR | 26
Statistical Analysis 1: Comparison: Carboplatin AUC-10; Test type: Other; Percentage = 45.0, 95% CI 2-sided [30.2 to 59.9]

3. Secondary Outcome: Overall Survival
Description: Survival status at 2 years after registration.
Time Frame: 2 years
Population: All participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Carboplatin AUC-10
Number analyzed (Participants) | 48
Participants
  Alive | 48
  Deceased | 0
Statistical Analysis 1: Comparison: Carboplatin AUC-10; Test type: Other; Percentage = 100, 95% CI 2-sided [92.6 to 100]

ADVERSE EVENTS:
Time Frame: Start of treatment until 30 days after last dose.
Arm/Group | Carboplatin AUC-10
All-Cause Mortality (participants affected / at risk) | 0/48
Serious Adverse Events (participants affected / at risk) | 12/48
Other Adverse Events (participants affected / at risk) | 47/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carboplatin AUC-10 (N=48)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (5)
Headache (Nervous system disorders) | 2 (2)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4)
Vomiting (Gastrointestinal disorders) | 2 (3)
Calculus bladder (Renal and urinary disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carboplatin AUC-10 (N=48)
Hypertension (Vascular disorders) | 1 (1)
Fatigue (General disorders) | 44 (111)
Pain (General disorders) | 6 (7)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (4)
Mood swings (Psychiatric disorders) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 1 (1)
Neutrophil count decreased (Investigations) | 34 (81)
Platelet count decreased (Investigations) | 28 (53)
Weight decreased (Investigations) | 1 (1)
Weight increased (Investigations) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 27 (49)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Neuropathy peripheral (Nervous system disorders) | 6 (7)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 13 (15)
Constipation (Gastrointestinal disorders) | 17 (26)
Diarrhoea (Gastrointestinal disorders) | 7 (11)
Gastritis (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 37 (70)
Stomatitis (Gastrointestinal disorders) | 16 (24)
Vomiting (Gastrointestinal disorders) | 14 (19)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (9)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 22 (38)
Infection (Infections and infestations) | 4 (5)
Neutropenic sepsis (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No PI may present data from his/her centre separately from the rest of the study results unless approved by the Trial Steering Committee and the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2017-08-31): https://cdn.clinicaltrials.gov/large-docs/16/NCT02272816/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-10): https://cdn.clinicaltrials.gov/large-docs/16/NCT02272816/SAP_001.pdf